CLINICAL TRIAL: NCT06555471
Title: A Single-arm, Phase II Exploratory Study of Sintilimab in Combination With Chemoradiotherapy in Elderly Patients With Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123323
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; S 1 (combination); Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy sintilimab combined with chemotherapy and radiotherapy (Experimental): Sintilimab (200mg iv q3w d1) combined with chemoradiation. The application of chemotherapy based on investigator's assessment, and if so, S-1 (po d1-d14，q3w； according to body surface area ：<1.5m^2 40mg/time；1.5~1.8m^2 50mg/time；>1.8m2 60mg/time) or capecitabine （1000mg/m2 Bid po d1-14，q3w，Reduce or discontinue depending on the condition of the subject.); Radiotherapy：once a day, five times a week, at a dose of 1.8-2 Gy/f, for a total of 45-50.4 Gy. Radiation therapy starts from the first cycle of Sintilimab Injection combined with chemotherapy.
  Maintenance therapy with sintilimab in combination with S-1 (po d1-d14，q3w； according to body surface area ：<1.5m^2 40mg/time；1.5~1.8m^2 50mg/time；>1.8m2 60mg/time) or capecitabine （1000mg/m2 Bid po d1-14，q3w，Reduce or discontinue depending on the condition of the subject.) up to 2 years.
  Interventions: Drug: Sintilimab; Drug: S-1; Drug: Capecitabine; Radiation: Extraperitoneal radiation therapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: 200mg iv q3w d1
Drug: S-1 — po d1-d14，q3w； according to body surface area ：<1.5m^2 40mg/time；1.5~1.8m^2 50mg/time；>1.8m2 60mg/time)
Drug: Capecitabine — 1000mg/m2 Bid po d1-14，q3w，Reduce or discontinue depending on the condition of the subject.
Radiation: Extraperitoneal radiation therapy — once a day, five times a week, at a dose of 1.8-2 Gy/f, for a total of 45-50.4 Gy. Radiation therapy starts from the first cycle of Sintilimab Injection combined with chemotherapy

SUMMARY:
This trial is a prospective, single-arm, single-centre, phase II clinical study to explore the efficacy and safety of sintilimab in combination with chemoradiation in subjects over 75 years of age with advanced gastric cancer.

Participants will:

Take sintilimab (200mg iv q3w d1) combined with chemoradiation. The application of chemotherapy based on investigator's assessment, and if so, S-1 (po d1-d14，q3w； according to body surface area ：<1.5m^2 40mg/time；1.5~1.8m^2 50mg/time；>1.8m2 60mg/time) or capecitabine （1000mg/m2 Bid po d1-14，q3w，Reduce or discontinue depending on the condition of the subject.); Radiotherapy：once a day, five times a week, at a dose of 1.8-2 Gy/f, for a total of 45-50.4 Gy. Radiation therapy starts from the first cycle of Sintilimab Injection combined with chemotherapy.

Subjects undergo an initial assessment of imaging, physical status, quality of life, and relevant laboratory tests after completion of 3 cycles of sintilimab combination chemotherapy, followed by assessments every 2 months, and after 3 full assessments, assessments every 3 months are initiated.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed locally advanced (T3-4N+M0) adenocarcinoma of the stomach and gastroesophageal junction (including signet ring cell carcinoma, mucinous adenocarcinoma, and hepatoid adenocarcinoma).
* HER-2 negative.
* Age ≥75 years.
* ECOG PS score of 0-2
* have at least one measurable lesion or assessable lesion according to RECIST v1.1.
* have adequate organ and bone marrow function as defined below:

  1. Haematology: absolute neutrophil count ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L; haemoglobin level ≥ 9.0 g/dL.
  2. Liver function: Serum total bilirubin (TBIL) ≤ 1.5× the upper limit of normal (ULN); for patients with liver metastases or a history/suspicion of Gilbert's syndrome (persistent or recurrent hyperbilirubinemia, primarily unconjugated hyperbilirubinemia without evidence of hemolysis or liver disease), TBIL ≤ 3× ULN; for patients without hepatocellular carcinoma (HCC) and liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN; for patients with HCC or liver metastases, ALT or AST ≤ 5× ULN.
  3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min; urine protein < 2+ on urine test paper.
  4. Coagulation function: activated partial thromboplastin time (APTT) and international normalised ratio (INR) ≤ 1.5×ULN.
  5. Cardiac enzyme profile within normal range
  6. Normal thyroid function, defined as thyrotropin (TSH) within normal range. If baseline TSH is outside the normal range, subjects may also be enrolled if total T3 (or FT3) and FT4 are within the normal range;
* expected survival time ≥ 12 weeks;
* Signed written informed consent and able to comply with protocol-specified visits and related procedures.

Exclusion Criteria:

* known endoscopic signs of active bleeding from the lesion.
* Near obstruction of the cardia and pylorus affecting feeding and gastric emptying, or impaired swallowing of tablets.
* Diagnosis of HER-2 positive adenocarcinoma of the stomach and gastro-oesophageal junction.
* Previous systemic therapy for advanced or metastatic adenocarcinoma of the stomach and gastro-oesophageal junction.
* Malignant disease other than gastric cancer diagnosed within 5 years prior to the first dose (excluding radically treated basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or radically resected carcinoma in situ);
* Currently being treated in an interventional clinical study or have been treated with another investigational drug or with an investigational device within 4 weeks prior to the first dose;
* Prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs targeting another stimulatory or synergistic inhibitor of T-cell receptors (e.g., CTLA-4, OX-40, CD137);
* active autoimmune disease requiring systemic therapy (e.g., use of disease-mitigating medications, glucocorticoids, or immunosuppressive agents) within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic therapy;
* are receiving systemic glucocorticoid therapy (excluding topical glucocorticosteroids by nasal spray, inhalation or other routes) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study; Note: Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are permitted;
* known for allogeneic organ transplantation (except corneal transplantation) or allogeneic haematopoietic stem cell transplantation;
* Known allergy (grade 3 or higher) to any monoclonal antibody or component of a chemotherapeutic drug (Tegretol/Capecitabine) preparation;
* has not fully recovered from toxicity and/or complications resulting from any intervention prior to initiation of therapy (i.e., ≤ Grade 1 or at baseline, excluding malaise or alopecia);
* known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positivity with a detectable HBV-DNA copy number greater than the upper limit of normal in the laboratory of the study centre); Note: Subjects with hepatitis B who meet the following criteria may also be enrolled:

  1. HBV viral load <1000 copies/ml (200 IU/ml) prior to the first dose, and subjects should receive anti-HBV therapy throughout the duration of study chemotherapeutic drug treatment to avoid viral reactivation;
  2. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required but close monitoring of viral reactivation is needed.
* Subjects with active HCV infection (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
* Live vaccination within 30 days prior to the first dose (Cycle 1, Day 1); NOTE: Receipt of injectable inactivated viral vaccine against seasonal influenza within 30 days prior to the first dose is permitted; however, receipt of live attenuated influenza vaccine administered intranasally is not permitted.
* the presence of any serious or uncontrolled systemic illness, such as:

  1. Significant and symptomatic uncontrollable abnormalities in rhythm, conduction or morphology of the resting electrocardiogram, such as complete left bundle branch block, heart block of degree II or greater, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) classification ≥ grade 2;
  3. Any arterial thrombosis, embolism or ischaemia such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischaemic attack within 6 months prior to enrolment for treatment;
  4. Unsatisfactory control of blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
  5. History of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to the first dose, or current clinically active interstitial lung disease;
  6. Active tuberculosis;
  7. Presence of active or uncontrolled infection requiring systemic therapy;
  8. Presence of clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver disease such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poorly controlled diabetes mellitus (fasting blood glucose (FBG) > 10 mmol/L);
  11. Urine routine suggestive of urinary protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g;
  12. Patients with mental disorders who are unable to co-operate with treatment;
* A medical history, evidence of disease, treatment, or abnormal laboratory test results that could potentially interfere with the study results or hinder the participant's full involvement in the research, or any other situation that the investigator deems unsuitable for inclusion in the study, or the investigator believes there are other potential risks that make the participant unsuitable for this study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  Proportion of participants in complete and partial remission
Disease control rate (DCR) | 24 months
  the proportion of patients who achieve tumor relief (PR+CR) and stable disease (SD)
Duration of response (DoR) | 24 months
  the time from onset of response to progression or death due to any reason, whichever occurs earlier
Progression free survival (PFS) | 24 months
  the time from initiation of treatment to the occurrence of disease progression or death, whichever occurs earlier.

SECONDARY OUTCOMES:
Overall survival | 24 months
  the time from initiation of treatment to death caused by any reasons.
Adverse reactions | 24 months
  According to the adverse event data of CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China